CLINICAL TRIAL: NCT06861816
Title: Fatigue, Ventilatory Functions, Physical Intolerance, and Life Quality in ESRD Adolescents: Response to Program of Walking With Dogs
Brief Title: Ventilatory Functions and Physical Intolerance in ESRD Adolescents: Response to Program of Walking With Dogs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00014233-25
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease; Hemolysis
MeSH Terms: conditions — Kidney Failure, Chronic; Hemolysis | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): End stage renal diseased adolescents (numbering twenty) will trained by incentive spirometer 30 min during the sessions of dialysis three applications weekly for 12 weeks. they will additionally walked freely with a dog 30 min three times weekly (in opposite days of hemodialysis). The duration of this trial will be 12 weeks.
  Interventions: Other: incentive spirometer and walking with dog
- group number 2 (Active Comparator): End stage renal diseased adolescents (numbering twenty) will trained by incentive spirometer 30 min during the sessions of dialysis three applications weekly for 12 weeks.
  Interventions: Other: training by incentive spirometer only

INTERVENTIONS:
Other: incentive spirometer and walking with dog — End stage renal diseased adolescents (numbering twenty) will trained by incentive spirometer 30 min during the sessions of dialysis three applications weekly for 12 weeks. they will additionally walked freely with a dog 30 min three times weekly (in opposite days of hemodialysis). The duration of this trial will be 12 weeks.
  Arms: group number 1
Other: training by incentive spirometer only — End stage renal diseased adolescents (numbering twenty) will trained by incentive spirometer 30 min during the sessions of dialysis three applications weekly for 12 weeks.
  Arms: group number 2

SUMMARY:
adolescents with chronic renal failure going on hemodialysis usually complain many problems including compromised ventilation, early fatigue, early physical intolerance, and bad life quality. incentive spirometer is highly recommended to improve these problems. also, walking program, especially walking with dog, can increase the benefits of incentive spirometer

DETAILED DESCRIPTION:
End stage renal diseased adolescents (numbering forty) will be grouped randomly to two random groups, twenty adolescents in group I or group II. Both groups will trained by incentive spirometer 30 min during the sessions of dialysis three applications weekly for 12 weeks. Group I will additionally walked freely with a dog 30 min three times weekly (in opposite days of hemodialysis). The duration of this trial will be 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* adolescents (forty) with ESRD
* patents on regular hemodiaysis

Exclusion Criteria:

* cardiac insult
* respiratory insult
* orthopedic problem
* liver insult

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
six minute walk testing | it will be measured after 12 weeks
  it is a physical capacity measure

SECONDARY OUTCOMES:
forced vital capacity | it will be measured after 12 weeks
  it is a pulmonary function test
forced expiratory volume at first second | it will be measured after 12 weeks
  it is a pulmonary function test
maximal inspiratory pressure | it will be measured after 12 weeks
  it is a test measures strength of inspiratory muscles
child health questionnaire (physical summary) | it will be measured after 12 weeks
  the parent form (50 questions) will used to measure quality of life
child health questionnaire (mental summary) | it will be measured after 12 weeks
  the parent form (50 questions) will used to measure quality of life
fatigue symptoms inventory | it will be measured after 12 weeks
  it is a questionnaire assesses fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt